CLINICAL TRIAL: NCT04121416
Title: Comparison of Effects of Oxycodone and Sufentanil on Cardiovascular Stress Induced by Tracheal Intubation in the Patients With Coronary Heart Disease Undergoing Major Noncardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Oxycodone VS Sufentanil
Record Dates: First submitted 2019-10-02; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular
Keywords: Oxycodone; Sufentanil; tracheal intubation
MeSH Terms: interventions — Oxycodone; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxycodone group (Experimental)
  Interventions: Drug: Oxycodone 10mg
- Sufentanil group (Experimental)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oxycodone 10mg — induction with 0.3mg/kg of oxycodone in general anesthesia
  Arms: Oxycodone group
Drug: Sufentanil — induction with 0.3 µg/kg of Sufentanil in general anesthesia
  Arms: Sufentanil group

SUMMARY:
To evaluate the effect of oxycodone and sufentanil in preventing cardiovascular responses to tracheal intubation in the patients with coronary heart disease (CHD).

DETAILED DESCRIPTION:
Laryngoscopy and tracheal intubation can provoke an increase of blood pressure (BP) and/or HR [1.2]. This hemodynamic stress may lead to an imbalance between myocardial oxygen consumption and supply and therefore induce myocardial ischemia, which may be endurable in the patients with normal cardiovascular condition but is potential harmful to the patients with coronary heart disease. Thus it is critical to attenuate the cardiovascular stress induced by laryngoscopy and endotracheal intubation in the high risk patients.

ELIGIBILITY:
Inclusion Criteria:

The coronary angiography from each patient showed that lesions exist in at least one main coronary artery

Exclusion Criteria:

a history of reactive airway disease, gastroesophageal reflux, morbid obesity, a known or predicted difficult airway

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
blood pressure(SBP)、diastolic blood pressure(DBP)、mean arterial pressure(MAP) | one second before anesthesia induction, the moment when tracheal catheter passes through glottis and at 1, 3, 5 min after tracheal intubation
  Under local anesthesia invasive artery line was put to the patients to monitor systolic blood pressure(SBP)、diastolic blood pressure(DBP)、mean arterial pressure(MAP)

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, Study Director — Shengjing Hospital
Locations (1):
- shengjing hospital of China medical university, Shenyang, Liaoning, China